CLINICAL TRIAL: NCT03072355
Title: Reliability and Validity of a Shoulder Fatigue Test Using Two Tools: Elastic Resistance and Isokinetic Dynamometer.
Brief Title: Reliability and Validity of a Shoulder Fatigue Test
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: São Paulo State University (Other)
Collaborators: Coordination for the Improvement of Higher Education Personnel (Other)
Responsible Party: Principal Investigator, Jaqueline Santos Silva, Master's Degree student, São Paulo State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: PP1
Record Dates: First submitted 2017-02-16; First posted 2017-03-07 (Actual); Last update posted 2017-11-09 (Actual); Status verified 2017-11

CONDITIONS: Healthy Volunteers
Keywords: fatigue; resistance test
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Elastic Band (Active Comparator): Perform the maximum of the possible repetition with a load of 50% of the 1RM (performing 1½ seconds in the concentric phase and 1½ seconds in the eccentric phase).
  Interventions: Other: Elastic Band
- Isokinetic dynamometer (Active Comparator): Realization of the maximum of the possible repetition to 50% of the MIVM in the speed of 60º / s for abduction and 500º / s in the return of the movement.
  Interventions: Other: Isokinetic dynamometer

INTERVENTIONS:
Other: Elastic Band — Localized muscle resistance test for shoulder
  Arms: Elastic Band
Other: Isokinetic dynamometer — Localized muscle resistance test for shoulder
  Arms: Isokinetic dynamometer

SUMMARY:
Introduction: The exercise performed with elastic tools has been appearing in the current scenario as a clinical tool because it presents advantages such as easy handling, low cost and safety. However, its use as an assessment tool, specifically for localized muscular resistance, is reduced and not standardized. In addition, there are no records of the physiological / neurofunctional effects of tests that use such a tool, since it allows a differentiated degree of prescription. Objective: To determine the reliability and reproducibility of a shoulder abduction resistance test in two tools, elastic tube and isokinetic dynamometer. In addition to analyzing the metabolic profile of both comparative order and targeting subsequent training prescription. Method: The study will consist of a sample of 30 participants and will be carried out in 2 stages, 15 participants will perform step 1 and the other 15 will perform step 2. The difference between the steps is the order of the tools used to perform the test . Each stage will consist of 5 sessions (Orientation, Familiarization 1 and 2, Test and Retest). During the test and retest sessions the physiological response of the test will be analyzed. In order to observe the response, will be analyzed the lactic anaerobic parameter (lactate concentration), allelic anaerobic (post-exercise oxygen uptake analysis - EPOC), aerobic parameter (VO2 values) and electromyographic measurements. Will be used the statistical package SPSS Statistics 22.0, Pearson's correlation and their respective confidence intervals will indicate the relationship between the numerical variables and multivariate models will be constructed by means of linear regression. The significance level of 5% will be adopted.

DETAILED DESCRIPTION:
Tests applied

1RM test The 1 RM test in the elastic band is based on the study by ANDERSEN et al. (2016). Elastic bands of the brand Theraband® CLX (Hygienic, Corporation, Akron, Ohio, USA) with a standard length of 1.47m, ranging from very low to very high strength (yellow, red, green, blue, black, silver, gold). Due to possible changes in the mechanical properties of elastic bands during the initial stretching cycles, all elastics will be pre-stretched 100 times.

Initially the research assistant will instruct the participants to sit on a chair, and place their feet together on the elastic band without shoes. Starting with the least elastic resistance (yellow), the research assistant will instruct the participants to perform a shoulder abduction of a unilateral (dominant) shoulder up to 90 ° and hold such a position for 3 seconds (statically). Thus, participants will have to perform the concentric contraction phase without the help of the research assistant before reaching the static test position. Through visual inspection, the search assistant will control the correct positioning of the movement. Two-minute intervals will be taught between resistance levels until it is not possible for the participant to reach and / or hold the position for 3 seconds. When there is a failure, two more attempts to reach and maintain the desired position will be accomplished. During the essay, the research assistant will provide verbal encouragement. The obtained torque will be calculated by a formula based on the study of ANDERSEN et al. (2016).

Isokinetic muscle strength test For the MVIC test, the participant will be seated with the dominant upper limb on the Biodex System Pro 4 isokinetic dynamometer (Biodex Medical System, Shirley-NY, USA). Prior to the test, the participant will undergo a warm-up consisting of 10 repetitions of concentric contraction of abduction-adduction of the shoulder at 180º / s throughout the range of motion. After the warm-up will be given a two-minute rest break to the start of the MVIC. The CIVM will be considered as the Of torque obtained between three 5 second repetitions of abduction, with the dominant upper limb positioned at 90º horizontal abduction of the shoulder. A two-minute interval between replicates will be administered in order to minimize possible fatigue effects. The participant will be instructed to perform their maximum power performance and will be verbally encouraged by the evaluator in each attempt made. Such protocol is based on the one used by BARONI et al., (2010) for lower limb.

Fatigue Resistance Test (TRF) TRF - Elastic Tube: To perform the fatigue resistance test on the elastic tube the participant will initially be positioned sitting on a chair with their feet together stepping on the elastic band without shoes. He will then perform a 20-second abduction-adduction heating of the shoulder from the neutral position to 90 °. The interval of 2 minutes will then be given to start the TRF. This will consist of performing the maximum of the possible repetition with a load of 50% of the 1RM (1½ second in the concentric phase and 1½ second in the eccentric phase).

TRF - Isokinetic Dynamometer: In order to perform the fatigue resistance test in the isokinetic dynamometer, the participant will initially be positioned with the dominant upper limb attached to the dynamometer by means of the apparatus itself. He will then perform a warm-up of 10 concentric contractions of abduction-adduction of the shoulder at 180º / s throughout the range of movement (0º to 90º). The interval of 2 minutes will then be given to start the TRF. This will consist of performing the maximum possible repetition at 50% of the MVIC at the rate of 60º / s for abduction and 500º / s at the return of the movement.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Male gender
* Aged between 18 and 30 years
* Agreement to participate through signed statement of informed consent

Exclusion Criteria:

* Be an alcoholic,
* Consume drugs,
* Consuming tobacco or anti-inflammatory medications in a chronic way,
* Anemia, an inflammatory process, diabetes, cardiovascular disease, and
* an episode of muscle-tendon or osteoarticular injury in the lower limbs and / or spine in the last six months.

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Males between the ages of 18 and 30, apparently healthy
Enrollment: 30 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2017-08-30 (Actual); Study Completion 2017-08-30 (Actual)

PRIMARY OUTCOMES:
Change in time values | 1 minute post test
  It will be divided into two stages. The 30 participants recruited will be randomized to perform the steps, 15 participants will perform step 1 and the other 15 participants will perform step 2. The difference between the participants is between the order of the procedures.
  In stage 1 the participants will perform 4 tests, the two tests initially with the device tube elastic the two ends with the isokinetic dynamometer, with 30 minutes interval between tests. For step 2, another 15 participants will perform the same procedures with the order of alternate tools. The change time values will be analyzed for reliability and reproducibility of the test.
Change in repetitions values | 1 minute post test
  It will be divided into two stages. The 30 participants recruited will be randomized to perform the steps, 15 participants will perform step 1 and the other 15 participants will perform step 2. The difference between the participants is between the order of the procedures.
  In stage 1 the participants will perform 4 tests, the two tests initially with the device tube elastic the two ends with the isokinetic dynamometer, with 30 minutes interval between tests. For step 2, another 15 participants will perform the same procedures with the order of alternate tools. The change on repetitions values will be analyzed for reliability and reproducibility of the test.

SECONDARY OUTCOMES:
Perception of effort | 1 minute post test 1, 1 minute post test 2, 1 minute post test 3, 1 minute post test 4.
  Evaluated through the OMNI Resistance Exercise Scale for Perceived Effort
Recovery Perception | 10 minute post test 1, 10 minute post test 2, 10 minute post test 3, 10 minute post test 4.
  Will be evaluated through the Likert Scale of Recovery Perception, with "one" corresponding to "not recovery" and 10 "fully recovery"
Psychological Questionnaire | Baseline
  Participants will be instructed to mark a dash on a visual analogue scale of 10 centimeters between two extremes, zero being "least possible" and 10 indicating "most possible" for each classification as previously described
Lactate concentration | baseline, 3, 5 and 7 minutes after the first test with both tools (Stage 1 and Stage 2)
  After 10 minutes of rest ([lacR]) and at moments 3, 5, and 7 minutes after the test (to determine the peak lactate concentration ([lacP]), 25 μl of arterialized blood of the patient will be collected in heparinized capillaries. Ear lobe, and discarded in plastic tubes (polyethylene) type Eppendorf (1.5 mL) containing 50 μl of sodium fluoride (NaF - 1%), for later lactacidemia analysis, performed in a lactomer.
Gas exchange | Immediately post test up to seven minutes post test
  Measurement of gas exchange throughout the test and up to 7 minutes at the end. Time-to-exhaustion analysis and post-exercise oxygen uptake (COPD).
Electromyographic measurements | 1 minute after the second test with both tools (Stage 1 and Stage 2)
  In addition to the variables related to the strength signal (FP,% AV, TC and TS), and the maximum amplitude in the EMG signal reached at the moment of the electrical stimulation, called M-Wave.

CONTACTS AND LOCATIONS:
Locations (1):
- Carlos Pastre, PhD, Presidente Prudente, Brazil

IPD SHARING:
Plan to Share IPD: No